CLINICAL TRIAL: NCT00845065
Title: A Phase 3 Safety and Efficacy Study of Boceprevir in Combination With Peginterferon Alfa-2a and Ribavirin in Subjects With Chronic Hepatitis C Genotype 1 Who Failed Prior Treatment With Peginterferon/Ribavirin
Brief Title: Boceprevir in Combination With Peginterferon Alfa-2a and Ribavirin in Participants With Chronic Hepatitis C Genotype 1 Who Failed Prior Treatment With Peginterferon/Ribavirin (Study P05685AM2)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P05685
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Results first posted 2012-02-02 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Control Arm) (Placebo Comparator): Peginterferon alfa-2a (180 μg/week subcutaneously [SC]) plus ribavirin (1000 to 1200 mg/day orally [PO]) for 4 weeks followed by placebo (800 mg three times a day [TID] PO, using placebo matching SCH 503034 200-mg capsules) + peginterferon alfa-2a 180 μg/week SC plus ribavirin 1000 to 1200 mg/day PO divided twice daily (BID) for 48 weeks with 24 weeks post-treatment follow-up.
  Interventions: Other: Placebo; Biological: Peginterferon alfa-2a; Drug: Ribavirin
- Arm 2 (Boceprevir Arm) (Experimental): Peginterferon alfa-2a (180 μg/week subcutaneously [SC]) plus ribavirin (1000 to 1200 mg/day orally [PO]) for 4 weeks followed by boceprevir (800 mg three times a day [TID] PO, using SCH 503034 200-mg capsules) + peginterferon alfa-2a 180 μg/week SC plus ribavirin 1000 to 1200 mg/day PO divided twice daily (BID) for 48 weeks
  with 24 weeks post-treatment follow-up.
  Interventions: Drug: Boceprevir; Biological: Peginterferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Boceprevir — 800 mg, using SCH 503034 200-mg capsules, three times a day (TID) orally (PO) for 48 weeks
  Other Names: SCH 503034
  Arms: Arm 2 (Boceprevir Arm)
Other: Placebo — 800 mg, using placebo matching SCH 503034 200-mg capsules, three times a day (TID) orally (PO) for 48 weeks
  Arms: Arm 1 (Control Arm)
Biological: Peginterferon alfa-2a — Peginterferon alfa-2a, pre-filled syringes, given 180 μg/week subcutaneously (SC) for 48 weeks
  Other Names: Pegasys®
Drug: Ribavirin — Ribavirin 200-mg capsules, weight-based dosing
  * <75 kg, 1000 mg/day orally (PO), divided twice daily (BID)
  * >=75 kg, 1200 mg/day PO, divided BID
  for 48 weeks
  Other Names: SCH 18908

SUMMARY:
Based on previous experience with peginterferon alfa-2b/ribavirin in combination with boceprevir, the combination with peginterferon alfa-

2a/ribavirin and boceprevir is expected to be safe and well tolerated. Given the wide utilization of both peginterferons and the clear benefit of the

addition of boceprevir to peginterferon alfa-2b/ribavirin, it is important to demonstrate the safety and efficacy of boceprevir in combination with

peginterferon alfa-2a/ribavirin.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a qualifying regimen defined as peginterferon alfa-2a/ribavirin or peginterferon alfa-2b/ribavirin for a minimum of 12 weeks.
* During the qualifying regimen, subjects must have either:

  * A documented undetectable Hepatitis C Virus-Ribonucleic Acid (HCV-RNA) within 30 days of the end-of-treatment and a subsequent detectable HCV-RNA during follow-up OR
  * A documented decline in HCV-RNA by >=2 log10 after 12 weeks of treatment.
* Subject must have previously documented chronic hepatitis C genotype 1 infection.
* Subject must have a liver biopsy with histology consistent with chronic hepatitis C infection and no other etiology.
* Subjects with bridging fibrosis or cirrhosis must have an ultrasound within 6 months with no findings suspicious for hepatocellular carcinoma (HCC).
* Subject must be >=18 years of age.
* Subject must weigh between 40 kg and 125 kg.
* Subject and subject's partner(s) must each agree to use acceptable methods of contraception.
* Subjects must be willing to give written informed consent.

Exclusion Criteria:

Subject will be excluded from entry if ANY of the criteria listed below are

met:

* Subjects known to be coinfected with the human immunodeficiency virus (HIV) or hepatitis B virus (hepatitis B surface antigen [HBsAg] positive) and/or demonstrating signs and symptoms consistent with co-infection.
* Subjects who required discontinuation of previous interferon or ribavirin regimen for an adverse event considered by the investigator to be possibly or probably related to ribavirin and/or interferon.
* Treatment with ribavirin within 90 days and any interferon alfa within 1 month of Screening.
* Treatment for hepatitis C with any investigational medication. Prior treatment with herbal remedies with known hepatotoxicity is exclusionary.
* Treatment with any investigational drug within 30 days of the randomization visit in this study.
* Participation in any other clinical trial within 30 days of randomization or intention to participate in another clinical trial during participation in this study.
* Evidence of decompensated liver disease.
* Diabetic and/or hypertensive subjects with clinically significant ocular examination findings.
* Pre-existing psychiatric condition(s).
* Clinical diagnosis of substance abuse.
* Any known pre-existing medical condition that could interfere with the subject's participation in and completion of the study.
* Evidence of active or suspected malignancy, or a history of malignancy, within the last 5 years (except adequately treated carcinoma in situ and basal cell carcinoma of the skin).
* Subjects who are pregnant or nursing. Subjects who intend to become pregnant during the study period. Male subjects with partners who are or who intend to become pregnant during the study period.
* Any other condition which, in the opinion of a physician, would make the subject unsuitable for enrollment or could interfere with the subject participating in and completing the study.
* Subjects who are part of the site personnel directly involved with this study.
* Subjects who are family members of the investigational study staff.
* Subjects who had a life-threatening serious adverse event (SAE) during the screening period.
* Subjects with a history of pancreatitis, except for one episode clearly secondary to gallstone.

Laboratory Exclusion Criteria:

* Hematologic, biochemical, and serologic criteria (growth factors may not be used to achieve study entry requirements):

  * Hemoglobin (Hgb) <12 g/dL for females and <13 g/dL for males
  * Neutrophils <1500/mm3 (blacks: <1200/mm3)
  * Platelets <100,000/mm3
  * Direct bilirubin >1.5 x upper limit of normal (ULN) of the laboratory reference range. Total bilirubin >1.6 mg/dL unless the subject has a history of Gilbert's disease. If Gilbert's disease is the proposed etiology, this must be documented in the subject's chart.
* Serum albumin < lower limit of normal (LLN) of laboratory reference range.
* Thyroid-stimulating hormone (TSH) >1.2 x ULN or <0.8 x LLN of laboratory reference range.
* Serum creatinine >ULN of the laboratory reference range.
* Serum glucose:

  * For subjects not previously diagnosed with diabetes mellitus:

    * >=140 mg/dL (nonfasting) unless hemoglobin A1c subtype (HbA1c) <=7% OR
    * >=100 mg/dL (fasting) unless HbA1c <=7%.
  * For subjects previously diagnosed with diabetes mellitus: HbA1c >8.5%.
* Prothrombin time/partial thromboplastin time (PT/PTT) values >10% above laboratory reference range.
* Anti-nuclear antibodies (ANA) >1:320.
* Alpha fetoprotein (AFP):

  * AFP >100 ng/mL OR
  * AFP 50 to 100 ng/mL requires a liver ultrasound and subjects with findings suspicious for HCC are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2009-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Flamm SL, Lawitz E, Jacobson I, Bourliere M, Hezode C, Vierling JM, Bacon BR, Niederau C, Sherman M, Goteti V, Sings HL, Barnard RO, Howe JA, Pedicone LD, Burroughs MH, Brass CA, Albrecht JK, Poordad F. Boceprevir with peginterferon alfa-2a-ribavirin is effective for previously treated chronic hepatitis C genotype 1 infection. Clin Gastroenterol Hepatol. 2013 Jan;11(1):81-87.e4; quiz e5. doi: 10.1016/j.cgh.2012.10.006. Epub 2012 Oct 10. PMID 23064222

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 202 participants were randomized but 1 participant was not treated.
Groups:
- PEG2a/Ribavirin: Peginterferon alfa-2a (PEG2a) (180 μg/week subcutaneously [SC]) plus ribavirin (1000 to 1200 mg/day orally [PO]) for 4 weeks followed by placebo (800 mg three times a day [TID] PO, using placebo matching SCH 503034 200-mg capsules) + PEG2a 180 μg/week SC plus ribavirin 1000 to 1200 mg/day PO divided twice daily (BID) for 48 weeks with 24 weeks post-treatment follow-up.
- Boceprevir/PEG2a/Ribavirin: PEG2a (180 μg/week SC) plus ribavirin (1000 to 1200 mg/day PO) for 4 weeks followed by boceprevir (800 mg TID PO, using SCH 503034 200-mg capsules) + PEG2a 180 μg/week SC plus ribavirin 1000 to 1200 mg/day PO divided BID for 48 weeks with 24 weeks post-treatment follow-up.
Period: Overall Study
Arm/Group | PEG2a/Ribavirin | Boceprevir/PEG2a/Ribavirin
Started | 67 | 134
Completed | 20 | 79
Not Completed | 47 | 55
Not completed — Adverse Event | 3 | 23
Not completed — Lack of Efficacy | 43 | 21
Not completed — Non-Medical Reasons | 1 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PEG2a/Ribavirin | Boceprevir/PEG2a/Ribavirin | Total
Number analyzed (Participants) | 67 | 134 | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (6.8) | 52.0 (7.2) | 52.5 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 37 | 61
  Male | 43 | 97 | 140

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virologic Response (SVR) Rate in Full Analysis Set (FAS) Population.
Description: SVR rate was the percentage of participants treated with at least one dose of study medication (PEG2a, Ribavirin, or Boceprevir/Placebo) who had achieved SVR. SVR was defined as undetectable Hepatitis C Virus-Ribonucleic Acid (HCV RNA).
Time Frame: Follow-up Week 24
Population: FAS Population: all randomized participants who received at least one dose of study medication (PEG2a, Ribavirin, or Boceprevir/Placebo). Follow-up (FU) Week (W) 12 value was Last Observation Carried Forward (LOCF), if last SVR value at or after FU W24 was not available.
Measure: Number; unit: Percentage of Participants
Arm/Group | PEG2a/Ribavirin | Boceprevir/PEG2a/Ribavirin
Number analyzed (Participants) | 67 | 134
Percentage of Participants | 20.9 | 64.2

2. Secondary Outcome: SVR Rate in the Modified Intent-to-Treat (mITT) Population
Description: SVR rate was the percentage of participants treated with at least one dose of study medication (Boceprevir/PEG2a/Ribavirin or PEG2a/Ribavirin). Participants who discontinued study drugs during the 4-week PEG2a/Ribavirin lead-in period were not included in the mITT population.
Time Frame: Follow-up Week 24
Population: mITT Population: all randomized participants who received at least one dose of study medication (Boceprevir/PEG2a/Ribavirin or PEG2a/Ribavirin). Participants who discontinued study drugs during the 4-week PEG2a/Ribavirin lead-in period were not included. FU W12 value was LOCF, if last SVR value at or after FU W24 was not available.
Measure: Number; unit: Percentage of Participants
Arm/Group | PEG2a/Ribavirin | Boceprevir/PEG2a/Ribavirin
Number analyzed (Participants) | 67 | 130
Percentage of Participants | 20.9 | 66.2

3. Secondary Outcome: Percentage of Participants With Early Virologic Response (EVR) Who Achieved SVR
Description: EVR was defined as the time to the first undectectable HCV-RNA result at Treatment Week (TW) 2, 4, 8, or 12. Participants with a detectable, but not quantifiable HCV-RNA result at TW 12 may have undergone retesting. Participants with a detectable result on retesting were to be discontinued per the 12-week futility rule. Participants with an undetectable result on retesting were allowed to continue on treatment, and the detectable but not quantifiable result was to be considered a false positive.
Time Frame: Day 1 to Treatment Week 12
Population: FAS Population
Measure: Number; unit: Percentage of Participants
Arm/Group | PEG2a/Ribavirin | Boceprevir/PEG2a/Ribavirin
Number analyzed (Participants) | 67 | 134
Percentage of Participants
  <=TW 4 (PEG2a N = 2, Boceprevir N = 3) | 50.0 | 100.0
  >TW 4 to TW 8 (PEG2a N = 7, Boceprevir N = 76) | 42.9 | 82.9
  >TW 8 to TW 12 (PEG2a N = 9, Boceprevir N = 22) | 88.9 | 68.2

4. Secondary Outcome: Number of Participants With Undetectable HCV-RNA at Follow-up Week 12
Time Frame: Follow-up Week 12
Population: FAS Population
Measure: Number; unit: Participants
Arm/Group | PEG2a/Ribavirin | Boceprevir/PEG2a/Ribavirin
Number analyzed (Participants) | 67 | 134
Participants | 12 | 87

5. Secondary Outcome: Mean Log Change From Baseline to TW 4 in Viral Load by Visit
Description: HCV-RNA levels were quantified using the Roche Cobas Taqman 1.0 assay; lower limit of detection of 15 international units [IU]/mL. Changes in HCV-RNA IU/ml were expressed on a log10 scale.
Time Frame: From Baseline to TW 4
Population: FAS Population
Measure: Mean (Standard Deviation); unit: log10 (IU/mL)
Arm/Group | PEG2a/Ribavirin | Boceprevir/PEG2a/Ribavirin
Number analyzed (Participants) | 67 | 134
log10 (IU/mL) | -2.44 (1.32) | -2.33 (1.34)

ADVERSE EVENTS:
Arm/Group | PEG2a/Ribavirin | Boceprevir/PEG2a/Ribavirin
Serious Adverse Events (participants affected / at risk) | 7/67 | 18/134
Other Adverse Events (participants affected / at risk) | 67/67 | 133/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG2a/Ribavirin (N=67) | Boceprevir/PEG2a/Ribavirin (N=134)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 1 (1)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
ASTHENIA (General disorders) | 0 (0) | 1 (1)
CHEST PAIN (General disorders) | 1 (1) | 0 (0)
IRRITABILITY (General disorders) | 1 (1) | 0 (0)
MULTI-ORGAN FAILURE (General disorders) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 0 (0) | 1 (2)
BRONCHITIS (Infections and infestations) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1)
CHLAMYDIAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 2 (2)
PNEUMONIA STAPHYLOCOCCAL (Infections and infestations) | 0 (0) | 1 (1)
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
UROSEPSIS (Infections and infestations) | 0 (0) | 1 (1)
FOREIGN BODY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
GUN SHOT WOUND (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
LETHARGY (Nervous system disorders) | 0 (0) | 1 (1)
NEURALGIA (Nervous system disorders) | 1 (1) | 0 (0)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 0 (0) | 2 (2)
ABNORMAL BEHAVIOUR (Psychiatric disorders) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 1 (1)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 1 (1)
RENAL COLIC (Renal and urinary disorders) | 1 (1) | 0 (0)
OSTEOTOMY (Surgical and medical procedures) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG2a/Ribavirin (N=67) | Boceprevir/PEG2a/Ribavirin (N=134)
ANAEMIA (Blood and lymphatic system disorders) | 22 (32) | 67 (119)
LEUKOPENIA (Blood and lymphatic system disorders) | 2 (3) | 20 (43)
NEUTROPENIA (Blood and lymphatic system disorders) | 12 (17) | 41 (89)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 4 (6) | 9 (12)
DRY EYE (Eye disorders) | 1 (1) | 9 (9)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 7 (8)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 4 (5) | 11 (12)
CONSTIPATION (Gastrointestinal disorders) | 5 (5) | 5 (5)
DIARRHOEA (Gastrointestinal disorders) | 5 (5) | 33 (38)
DRY MOUTH (Gastrointestinal disorders) | 2 (2) | 7 (7)
DYSPEPSIA (Gastrointestinal disorders) | 3 (3) | 10 (11)
NAUSEA (Gastrointestinal disorders) | 18 (19) | 52 (60)
VOMITING (Gastrointestinal disorders) | 0 (0) | 16 (21)
ASTHENIA (General disorders) | 12 (15) | 29 (47)
CHILLS (General disorders) | 8 (8) | 14 (24)
FATIGUE (General disorders) | 36 (43) | 67 (80)
INFLUENZA LIKE ILLNESS (General disorders) | 18 (18) | 35 (37)
INJECTION SITE ERYTHEMA (General disorders) | 4 (4) | 9 (9)
IRRITABILITY (General disorders) | 16 (17) | 29 (34)
OEDEMA PERIPHERAL (General disorders) | 3 (3) | 7 (8)
PAIN (General disorders) | 2 (2) | 9 (10)
PYREXIA (General disorders) | 8 (8) | 18 (39)
INFLUENZA (Infections and infestations) | 0 (0) | 8 (8)
WEIGHT DECREASED (Investigations) | 4 (4) | 11 (12)
DECREASED APPETITE (Metabolism and nutrition disorders) | 12 (12) | 27 (28)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 12 (15) | 16 (22)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 (6) | 10 (12)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 5 (7) | 14 (16)
MYALGIA (Musculoskeletal and connective tissue disorders) | 5 (5) | 25 (32)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 7 (8)
DISTURBANCE IN ATTENTION (Nervous system disorders) | 4 (4) | 8 (9)
DIZZINESS (Nervous system disorders) | 10 (10) | 17 (19)
DYSGEUSIA (Nervous system disorders) | 10 (10) | 52 (53)
HEADACHE (Nervous system disorders) | 21 (25) | 37 (46)
ANXIETY (Psychiatric disorders) | 9 (9) | 16 (18)
DEPRESSION (Psychiatric disorders) | 6 (7) | 22 (28)
INSOMNIA (Psychiatric disorders) | 20 (21) | 32 (36)
SLEEP DISORDER (Psychiatric disorders) | 3 (4) | 15 (16)
COUGH (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 26 (32)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 26 (28)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 13 (16)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 13 (15)
ALOPECIA (Skin and subcutaneous tissue disorders) | 5 (5) | 22 (24)
DRY SKIN (Skin and subcutaneous tissue disorders) | 11 (13) | 20 (22)
PRURITUS (Skin and subcutaneous tissue disorders) | 8 (9) | 18 (23)
RASH (Skin and subcutaneous tissue disorders) | 5 (5) | 31 (37)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator agrees not to present any interim results of study without prior written consent of sponsor. Investigator agrees to provide sponsor 45 days prior to submission publication, review copies of abstracts/manuscripts that report any results of the study. Sponsor shall have the right to review/comment on data analysis. If parties disagree investigator agrees to meet with sponsor's representatives at clinical study site for purpose of making good faith efforts to resolve any such issues.